CLINICAL TRIAL: NCT03148314
Title: Home-Based Extended Low Dose Buccal Misoprostol Versus Hospital-Based Standard Vaginal Dose In Management Of First Trimester Missed Abortion.
Brief Title: Vaginal Misoprostol In Management Of First Trimester Missed Abortion.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohammed Khairy Ali, Lecturer of obstetrics and gynecology, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VMIS
Record Dates: First submitted 2017-05-08; First posted 2017-05-11 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Abortion, Missed
MeSH Terms: conditions — Abortion, Missed

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- hospital- based vaginal misoprostol (Active Comparator): hospital- based vaginal misoprostol
  Interventions: Drug: vaginal misoprostol
- extended low dose oral misoprostol (Active Comparator): extended low dose oral misoprostol
  Interventions: Drug: buccal/sublingual misoprostol

INTERVENTIONS:
Drug: vaginal misoprostol — (800µgm.x 2 doses 3 hours).
  Other Names: buccal/sublingual misoprostol
  Arms: hospital- based vaginal misoprostol
Drug: buccal/sublingual misoprostol — 200 µgm.x4 hrs.x 6 doses
  Other Names: vaginal misoprostol
  Arms: extended low dose oral misoprostol

SUMMARY:
The world health organization defined abortion or miscarriage as : the expulsion or extraction from its mother of a fetus or an embryo weighting 500 grams or less ,or any other wise product of gestation of any weight irrespective of gestational age and weather or not there is evidence of life and weather or not the abortion was spontaneous or induced Miscarriage is the most common complication of pregnancy occurring in 10-20% of clinically recognized pregnancies (Bag. It is estimated that around 40% of early pregnancies result in miscarriage. A large majority of those are lost before the menstrual period is missed. More than 80%of abortions occur in first 12 weeks of pregnancy, and the rate decrease there after For clinical purposes: abortion is subdivided into: threatened abortion, inevitable abortion, incomplete abortion ,missed abortion ,septic abortion ,and recurrent abortion

ELIGIBILITY:
Inclusion Criteria:

* single dead fetus up-to 12 weeks.
* no low lying placenta
* no scarred uterus
* no or mild bleeding
* no evidence of infection
* accepting to participate in the study.

Exclusion Criteria:

* Advanced hepatic diseases .
* Suspected molar pregnancy
* Ectopic pregnancy or pregnancy of unknown location
* Haemodynamically unstable with significant anaemia ie Hb<10
* Uncontrolled severe asthma
* Chronic adrenal failure
* Known or suspected heart disease
* Glaucoma
* Haemoglobinopathies
* Haemorrhagic disorders and anti-coagulation therapy (aspirin accepted)
* Adrenal suppression and long term glucocorticoid therapy (may require corticosteroid)
* Patient living in remote areas with difficulty in accessing hospital

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 140 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2018-06-01 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with complete abortion (success rate). | 1 week

SECONDARY OUTCOMES:
Number of misoprostol doses | 1 week
induction-abortion time | 1 week

CONTACTS AND LOCATIONS:
Locations (1):
- Women Health Hospital - Assiut university, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ghosh J, Papadopoulou A, Devall AJ, Jeffery HC, Beeson LE, Do V, Price MJ, Tobias A, Tuncalp O, Lavelanet A, Gulmezoglu AM, Coomarasamy A, Gallos ID. Methods for managing miscarriage: a network meta-analysis. Cochrane Database Syst Rev. 2021 Jun 1;6(6):CD012602. doi: 10.1002/14651858.CD012602.pub2. PMID 34061352